CLINICAL TRIAL: NCT06416449
Title: The Effect of Kinesio Taping on Balance, Agility, and Jumping Performance in Adolescent Basketball Players Aged 12-18.
Brief Title: The Impact of Kinesio Taping on Balance, Agility, and Jumping in Adolescent Basketball Players Aged 12-18.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, AYCAN ÇAKMAK REYHAN, Principal Investigator, Istanbul Bilgi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: İstanbulBUuuuu
Record Dates: First submitted 2024-04-17; First posted 2024-05-16 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Balance; Jumping Performance; Agility Test
Keywords: kinesio taping, , balance, agility and jumping performance; basketball players; balance, agility; jumping performance

STUDY DESIGN:
Intervention Model Description: We'll assess balance, agility, and jumping. Tests include Star Balance Test, T-Agility Test, and Vertical Jump Test. In Star Balance, lines are drawn on the ground, the individual stands on one foot, reaching out with the other to touch lines. In T-Agility, a course is set, and time is recorded. The Vertical Jump Test measures the highest point reached against a wall-mounted ruler. Kinesio tape, allowing 55-60% elongation, will be used. Tests are conducted both with and without tape, with rest intervals.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Experimental): the Star Balance Test, lines are drawn on the ground. The individual stands on their dominant foot and reaches out with the tip of the contralateral foot to touch these lines, and points are recorded.
  the T-Agility Test, a course is set up, and the participant is asked to complete it as quickly as possible, with time being recorded.
  the Vertical Jump Test, the individual is asked to jump as high as possible against a wall-mounted ruler, and the highest point reached is recorded.
  The Kinesio tape used in the study is designed to reflect the characteristics of the skin and allow for approximately 55-60% elongation of its original length. These tests are first conducted without Kinesio tape and then repeated with Kinesio tape applied. Rest intervals are provided between tests.
  Interventions: Other: kinesiotape application

INTERVENTIONS:
Other: kinesiotape application — In the Star Balance Test, lines are drawn on the ground. The individual stands on their dominant foot and reaches out with the tip of the contralateral foot to touch these lines, and points are recorded. For the T-Agility Test, a course is set up, and the participant is asked to complete it as quickly as possible, with time being recorded.
  As implied by its name, cones are placed in a T-shape for the T-Agility Test, and the individual is required to touch the cones and return to the starting point as quickly as possible. In the Vertical Jump Test, the individual is asked to jump as high as possible against a wall-mounted ruler, and the highest point reached is recorded. The Kinesio tape used in the study is designed to reflect the characteristics of the skin and allow for approximately 55-60% elongation of its original length. These tests are first conducted without Kinesio tape and then repeated with Kinesio tape applied. Rest intervals are provided between tests.

SUMMARY:
In this study involving adolescent individuals who play basketball, we will investigate the effect of kinesio taping. Kinesio taping can be applied with appropriate technique and tension to reduce pain, swelling, and muscle spasms, as well as to correct mechanical issues. In this study, researchers will apply kinesio taping to the ankle and knee and thes assess its impact on balance, agility, and jumping performance through various tests. Specifically, researchers will conduct the star balance test for balance, the T-test for agility, and the vertical jump test for jumping performance. researchers plan to carry out this research with 30 participants at the Dev Ataşehir Sports Club to gather the necessary data.

DETAILED DESCRIPTION:
Basketball is a physically demanding and high-paced sport that requires balance, strength, stability, and agility. Kinesio taping, a method commonly used in athlete health where physiotherapists are involved, will be examined for its effect on the lower extremities of young basketball players. Kinesio tape allows for approximately 50-60% elongation of its own length and has a thickness similar to that of the epidermis layer of the skin. It can be applied with appropriate technique and tension to reduce pain, swelling, and muscle spasms, as well as to correct mechanical issues. In this study, researchers aimed to investigate the effect of kinesio taping on adolescent male basketball players. Kinesio taping will be applied to two different areas: the ankle and knee regions. The overall goal of this application is to increase stability and balance. The results of the applied tests will be evaluated. The effects of kinesio taping on balance, agility, and jumping performance in basketball players will be examined. In the research, parameters of balance, agility, and jumping performance will be examined. Researchers have specific tests for these parameters, including the Star Balance Test for balance, the T-Agility Test for agility, and the Vertical Jump Test for jumping performance. In the Star Balance Test, lines are drawn on the ground. The individual stands on their dominant foot and reaches out with the tip of the contralateral foot to touch these lines, and points are recorded. In the T-Agility Test, a course is set up, and the participant is asked to complete it as quickly as possible, with time being recorded.

As implied by its name, cones are placed in a T-shape for the T-Agility Test, and the individual is required to touch the cones and return to the starting point as quickly as possible. In the Vertical Jump Test, the individual is asked to jump as high as possible against a wall-mounted ruler, and the highest point reached is recorded. The Kinesio tape used in the study is designed to reflect the characteristics of the skin and allow for approximately 55-60% elongation of its original length. These tests are first conducted without Kinesio tape and then repeated with Kinesio tape applied. Rest intervals are provided between tests.

All participants will be asked to fill out a sociodemographic form and a consent form

ELIGIBILITY:
Inclusion Criteria:

* Participants must be athletes. They must have been engaged in sports for at least 1 year. Only male individuals will be included. Male individuals aged between 12 and 18 will be included.

Exclusion Criteria:

* Participants must not have experienced ankle or knee injuries in the last 3 months.

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The Star Balance Test | baseline and Immediately after application
  The Star Balance Test" is a method used to evaluate balance and stability. It involves standing on one leg at the center of a star-shaped platform. This test assesses an individual's ability to maintain balance, providing insight into proprioception and coordination skills. It's commonly used in sports medicine and rehabilitation
T-Agility Test | baseline and Immediately after application
  The T-Agility Test is a fitness assessment that evaluates agility, speed, and change-of-direction ability. Participants sprint forward, laterally shuffle to touch markers on each side, and return to the starting point. It's commonly used in sports training and fitness testing to measure quick directional changes.
Vertical Jump Test | baseline and Immediately after application
  The Vertical Jump Test measures lower body power and explosiveness. Participants jump vertically, reaching upwards to mark their maximum height. It's widely used in sports and fitness testing for assessing performance and tailoring training programs.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)